CLINICAL TRIAL: NCT03587688
Title: Registry for Mitral Valve Surgery at Department of Cardiac Surgery University Hospital of Basel/ Switzerland
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-00246,ch18Grapow
Record Dates: First submitted 2018-07-03; First posted 2018-07-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Mitral Valve Disease; Mitral Valve Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: mitral valve surgery — pre-, intra- and postoperative data on patients undergoing mitral valve surgery at the Department for Cardiac Surgery of Universitätsspital Basel/ Switzerland since 2009

SUMMARY:
A registry is installed to collect (pre-, intra- and postoperative) data on patients undergoing mitral valve surgery at the Department for Cardiac Surgery of Universitätsspital Basel/ Switzerland since 2009. Retrospective data (since 2009) as well as prospective data are included in this ongoing registry to analyse the development of mitral valve surgery at the Department of Cardiac Surgery University Hospital of Basel/ Switzerland.

ELIGIBILITY:
Inclusion Criteria:

- patients undergoing mitral valve surgery at the Department for Cardiac Surgery of Universitätsspital Basel/ Switzerland since 2009

Exclusion Criteria:

- patients refusing consent for data use

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients undergoing mitral valve surgery at the Department for Cardiac Surgery of Universitätsspital Basel/ Switzerland since 2009
Sampling Method: Probability Sample
Enrollment: 701 (Actual)
Dates: Start 2018-04-28 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
correlation between technique of mitral valve surgery and postoperative mitral valve pressure gradient | 4 weeks post surgery
  correlation between technique of mitral valve surgery and postoperative mitral valve pressure gradient

CONTACTS AND LOCATIONS:
Overall Officials: Martin Grapow, Prof. MD, Principal Investigator — University Hospital Basel, CH-4031 Basel
Locations (1):
- Herzchirurgie University Hospital Basel, Basel, Switzerland